CLINICAL TRIAL: NCT07094308
Title: Improving Outcomes in Chronic Intestinal Failure Using the ECHO Model: The LIFT-ECHO Last Mile Project
Brief Title: The LIFT-ECHO Last Mile Project
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Rhode Island Hospital (Other); The New York Academy of Medicine (Other); University of Utah (Other); London School of Economics and Political Science (Other)
Responsible Party: Principal Investigator, Kishore Iyer, Professor of Surgery, Pediatrics & Global Health, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY-23-00728
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Intestinal Failure
MeSH Terms: conditions — Intestinal Failure | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physicians with No Tele-Mentoring then with Tele-Mentoring (Active Comparator): Dyads consisting of a prescribing physician and one or more of their patients receiving parenteral nutrition (PN). Physicians in this arm will be invited to participate but would not yet have received the Tele-Mentoring (LIFT-ECHO) focused on the management of chronic intestinal failure. Patients of these physicians will be followed for a baseline period of 6 months (Control period) to assess evolution in clinical outcomes and patient-reported quality of life.
  Interventions: Behavioral: Learn Intestinal Failure Tele-ECHO Program; Behavioral: Standard of Care
- Physicians with Tele-Mentoring after No Tele-Mentoring (Experimental): Dyads consisting of a prescribing physician and one or more of their patients receiving parenteral nutrition (PN). Physicians in this arm will participate in the LIFT-ECHO program. After patients complete a baseline period of 6 months (Control period), their physician receives the intervention (LIFT-ECHO).
  Interventions: Behavioral: Learn Intestinal Failure Tele-ECHO Program; Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Learn Intestinal Failure Tele-ECHO Program — LIFT-ECHO (Learn Intestinal Failure Tele-ECHO) is a virtual tele-education program designed to improve the knowledge and clinical decision-making of non-specialist clinicians managing patients with chronic intestinal failure (CIF) on parenteral nutrition (PN). The intervention consists of eight 60-90-minute sessions delivered over 2-4 months. Each session includes the presentation of anonymized real-world CIF cases and a didactic lecture by an expert in intestinal rehabilitation. Participating physicians may also complete baseline and follow-up surveys, and optionally participate in focus groups or appreciative inquiry workshops.
  Other Names: LIFT-ECHO
Behavioral: Standard of Care — Participants will receive routine clinical care for chronic intestinal failure from their usual providers. No additional educational programming or intervention is delivered during this period.

SUMMARY:
This is a multi-site research study to evaluate the efficacy and effectiveness of the LIFT-ECHO program to improve clinical outcomes in patients and improve patient reported quality of life (PRQOL). LIFT-ECHO (Learn Intestinal Failure Tele-ECHO) is a tele-health learning program whereby non-specialist clinicians meet with and learn from CIF specialist teams with the goal of improving the knowledge of CIF. LIFT-ECHO sessions consist of group discussion of anonymized real-world patient cases, followed by a didactic presentation from an expert in intestinal failure. Sessions are held twice a month and last 60-90 minutes. The study will proceed in three distinct phases, correlating with Project Aims. During phase 1 (Aim 1), an intestinal failure disease activity index (IF-DAI) will be developed as a measure of short- to medium-term clinical activity in CIF patients; this phase will be undertaken through Delphi Rounds. During Phase 2 (corresponding to project Aim 2), the researchers will evaluate the impact of physician participation in LIFT-ECHO on patients with CIF on PN. Lastly, Phase 3, corresponding to Aim 3 will be the dissemination of LIFT-ECHO nationally. For Phase 2, the researchers had originally proposed that patients and physicians will be recruited from the records of Optum Home Infusion services. Patient reported quality of life and clinical status will be assessed using surveys at baseline. Physicians will then be invited to participate in a module of LIFT-ECHO consisting of 8 one- hour-long sessions held over the course of 2-4 months. Patients will then be followed for 12 months to assess if physician participation in LIFT-ECHO improves patient reported quality of life and/or treatment efficacy and effectiveness. The main procedures for physician participants in the study include: completion of baseline and monthly surveys, possible participation in an appreciative inquiry workshop and possible participation in a focus group discussion, optional, but encouraged, participation in LIFT-ECHO. The main procedures for patient participants include: completion of surveys at baseline, participation in 12 monthly follow-up phone calls with a study team member. The proposed trial has a total length of 34 months.

DETAILED DESCRIPTION:
The proposed trial includes baseline and post-LIFT-ECHO and consists of a minimum 150 clusters - defined as the unit of randomization, each representing one physician, with at least 1-n nested patients with CIF (>300 patients). The study comprises a minimum of four pre-defined sequences, with the exact number of sequences being based on the total number of physicians recruited for the trial. To perform the trial, all participating physicians are randomly selected to transition from the control group to the LIFT-ECHO intervention group, using a computer-generated algorithm (e.g., nQuery Advisor). Once a cluster crosses over to the intervention, it will remain exposed to the intervention for the remaining duration of the study, even if the actual LIFT-ECHO Module is only for 2 months. After each cluster has crossed over and transitioned to the intervention, there will be a 12-month period of follow-up during which all patients will remain treated. The trial requires that all participating physicians begin the control phase of the trial when the data collection period begins for patients and physicians (baseline period of 6 months).

ELIGIBILITY:
Inclusion Criteria:

* CIF patient participants must meet the following criteria in order to be considered eligible for participation:

  * Individuals of adult age (18 years or older), including pregnant women or Individuals of age > 5 years with parental consent and patient assent.
  * Diagnosis of chronic intestinal failure (ie. on PN >6 months with no malignancy, no HIV and a malabsorption or post-surgical diagnosis)
  * Currently receiving PN from a homecare infusion service company
* Physician Inclusion Criteria:

  * Physician participants must meet the following criteria in order to be considered eligible for participation:

    * Individuals of adult age (18 years or older), including pregnant women
    * Hold an MD or DO degree
    * Be a licensed physician prescriber with a homecare infusion service company

Exclusion Criteria:

* Participants meeting one or more of the following criteria will be excluded from participation:

  * Adults unable to consent (individuals with impaired decision-making capacity)
  * Prisoners
  * Children > 5 years who dissent

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Quality of Life (PRQOL) Score | Baseline, 6 months, and 12 months
  Patient-reported quality of life will be measured using the HPN-PROQ, a validated instrument designed for individuals receiving home parenteral nutrition (HPN). The total score ranges from 0 to 100, with higher scores indicating better quality of life. Subscales include physical health, emotional well-being, social functioning, and treatment burden, each also scored from 0 to 100, where higher scores indicate more favorable outcomes

SECONDARY OUTCOMES:
Intestinal Failure Disease Activity Index (IF-DAI) Score | Baseline through 12 months
  Intestinal Failure-Disease Activity Index (IF-DAI) is a composite clinical index to quantify disease activity in patients with chronic intestinal failure, incorporating weighted indicators such as central line infections, liver dysfunction, hospitalization, and GI-related procedures. Scores will be scaled such that higher scores indicate greater disease activity (i.e., worse clinical status). The IF-DAI is still in development and the minimum and maximum scores are to be determined.
Number of physicians recruited | Baseline through 12 months
  Feasibility of the LIFT-ECHO intervention will be assessed using physician recruitment.
Proportion of total physicians who completed at least 4 ECHO sessions | Baseline through 12 months
  Feasibility of the LIFT-ECHO intervention will be assessed using retention rates. Retention rate will be reported as proportion of total physicians who completed at least 4 ECHO sessions (Retention Rate = [Total # of physician subjects consented / Total # of physicians subjects who attended ≥4 ECHO sessions] *100).
Attendance number at ECHO sessions | Baseline through 12 months
  Feasibility of the LIFT-ECHO intervention will be assessed using physician attendance at ECHO sessions. Higher participation will indicate greater feasibility.
Number of ECHO sessions completed | Baseline through 12 months
  Feasibility of the LIFT-ECHO intervention will be assessed using completion of ECHO sessions. Higher completion rates will indicate greater feasibility.
Physician Satisfaction Scale | Post-intervention (within 1 month after final ECHO session)
  Acceptability will be measured using physician satisfaction. Survey is a Likert-scale with items scored from 1 (strongly disagree) to 5 (strongly agree) assessing satisfaction. Total scale is 1-5, with higher scores will indicate greater acceptability of the intervention.
Perceived usefulness Scale | Post-intervention (within 1 month after final ECHO session)
  Acceptability will be measured using perceived usefulness. Survey is a Likert-scale with items scored from 1 (strongly disagree) to 5 (strongly agree) assessing perceived usefulness. Total scale is 1-5, with higher scores will indicate greater acceptability of the intervention.
Likelihood of recommending LIFT-ECHO | Post-intervention (within 1 month after final ECHO session)
  Acceptability will be measured using likelihood of recommending LIFT-ECHO to others. Survey is a Likert-scale with items scored from 1 (strongly disagree) to 5 (strongly agree) assessing likelihood of recommending LIFT-ECHO to others. Total scale is 1-5, with higher scores will indicate greater acceptability of the intervention.
Physician Participation Rate | Baseline through 12 months
  Participation rate will be measured by tracking the number of physicians who enroll in the LIFT-ECHO program and attend at least one session. The proportion of participants who choose to participate, expressed as a percentage. Higher percentages indicate greater engagement with the program.
Number of Emergency Room Visits | Monthly up to 12 months
  Number of ER visits reported monthly by patients.
Number of Hospital Admissions | Monthly up to 12 months
  Number of hospital admissions reported monthly by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Iyer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (4):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - New York Academy of Medicine (NYAM), New York, New York
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Utah, Salt Lake City, Utah
- London School of Economics and Political Science, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Specify Other Mechanism Proposals should be submitted to marjorie.nisenholtz@mountsinai.org. All requests will be reviewed for methodological soundness and alignment with original consent and privacy protections. Approved users will be required to sign a Data Use Agreement. Data will be hosted on a secure institutional repository for a minimum of 5 years following publication.